CLINICAL TRIAL: NCT03138057
Title: Comparison of Fecal Digestive Enzymes in Infant Aged Between 0-1 Years Old
Brief Title: BM Characterization Pilot
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-17-02
Record Dates: First submitted 2017-04-20; First posted 2017-05-03 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Diaper Rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, pilot study to explore the relationship between an infant's nutrition, skin and stool composition at different ages.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0-12 months

Exclusion Criteria:

* Formula Fed
* Use of topical or oral antibiotics or antifungals within the past 4 weeks

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample of male and female infants who are not formula fed
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To determine enzymes in infant stools | approximately 1 week
  enzyme levels and activity of infant stools

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bargen, MD, Principal Investigator — Midwest Children's Health Research Institute
Locations (1):
- Midwest Children's Health Research Institute, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No